CLINICAL TRIAL: NCT04548830
Title: Safety of Transbronchial Cryobiopsy in a Cancer Population
Brief Title: Safety of Lung Cryobiopsy in People With Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-374
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer
Keywords: Cryobiopsy; 20-374
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single center investigator initiated study for patients who display indeterminant pulmonary nodules and diffuse parenchymal lung disease on CT chest imaging who have been referred to the Pulmonary service.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transbronchial cryobiopsy (Experimental): All study participants will undergo transbronchial biopsies via our proposed standardized cryo-biopsy protocol in place of the traditional forceps transbronchial biopsy that is typically used at MSK.
  Interventions: Procedure: Transbronchial cryobiopsy

INTERVENTIONS:
Procedure: Transbronchial cryobiopsy — After enrollment, and pre-treatment procedures are complete, patients will undergo flexible bronchoscopy with a therapeutic bronchoscope under general anesthesia via an advanced airway at Memorial Hospital in an inpatient or outpatient setting.

SUMMARY:
The purpose of this study is to find out whether a biopsy technique called transbronchial cryobiopsy (TBCB) is a safe alternative to the standard biopsy procedure (transbronchial forceps biopsy; TBFB). The study researchers think that TBCB may provide better biopsy samples to help diagnose lung disease.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater
* Patients with known or suspected diagnosis of cancer and indeterminant pulmonary nodules or diffuse parenchymal lung disease with non-diagnostic clinical profiles for whom a lung biopsy is deemed useful for diagnosis.

Exclusion Criteria:

* Patients with pulse oximetry less than 92% on oxygen delivery up to 2 L nasal cannula.
* Uncorrectable coagulopathy defined as:

  * Platelet count <50,000 x 10^9/L or
  * prothrombin time international normalized ratio >1.5
* Known pulmonary hypertension or echocardiographic pulmonary artery systolic pressure >50mmHg
* A secure diagnosis based on clinical and high-resolution CT scan data.
* Antiplatelet therapy that cannot be held for more than 5 days.
* Any patient deemed unfit to undergo bronchoscopy by the proceduralist
* Female patients with a positive pregnancy test within 30 days of the planned study procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Post Cryobiopsy complications | 2 years
  will be graded according to Common Terminology Criteria for Adverse Events version 5 (CTCAE v5)

CONTACTS AND LOCATIONS:
Overall Officials: Or Kalchiem-Dekel, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Husta BC, Ganjaei KG, Knezevic A, Aly RG, Fanaroff R, Lee RP, Bott MJ, Oberg CL, Travis WD, Chawla M, Kalchiem-Dekel O. A Prospective Study of Safety and the Incremental Diagnostic Value of Transbronchial Cryobiopsy Incorporated into Robotic-Assisted Bronchoscopy in a Cancer Population. Lung. 2025 Dec 18;204(1):1. doi: 10.1007/s00408-025-00863-x. PMID 41413664
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm